CLINICAL TRIAL: NCT03542864
Title: Medical Supervised Duodenal-Enteral Feeding for Overweight, Obesity and Increased Body Fat Percentage Treatment
Brief Title: Medical Supervised Duodenal-Enteral Feeding Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BiomediKcal (Other)
Collaborators: University of Alicante (Other); Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Isaac Kuzmar, MD, MBT, MsCN, PhD, Principal Investigator, BiomediKcal
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCE26418
Record Dates: First submitted 2018-04-26; First posted 2018-05-31 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Obesity, Visceral; Overweight and Obesity; Body Fat Disorder; Feeding and Eating Disorders; Hormone Disturbance; Weight Loss
Keywords: obesity; overweight; fat percentage; body fat; enteral feeding; fat loss
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Overweight; Feeding and Eating Disorders; Endocrine System Diseases; Weight Loss | interventions — Helio Progress

STUDY DESIGN:
Intervention Model Description: Duodenal-Enteral medical supervised feeding response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nasogastroduodenal Protocol (Experimental): Evaluation of a protocol for the treatment of excess body fat through duodenal nutrition
  Interventions: Dietary Supplement: Nasogastroduodenal Protocol
- Controls (Active Comparator): Change from Baseline Body Composition values at 1 and 3 months
  Interventions: Other: Control
- Data analysis (Other): Analysis and publication of data
  Interventions: Other: Data analysis

INTERVENTIONS:
Dietary Supplement: Nasogastroduodenal Protocol — Complete nutrition (carbohydrates, lipids, proteins, vitamins, oligoelements)
  Other Names: Medical-Clinical-Nutrition assessment
  Arms: Nasogastroduodenal Protocol
Other: Control — Progress registration of body composition values
  Other Names: Progress
  Arms: Controls
Other: Data analysis — Statistical analysis of all data
  Other Names: Statistics
  Arms: Data analysis

SUMMARY:
Medical Supervised Duodenal-Enteral Feeding for Overweight, Obesity and Increased Body Fat Percentage Treatment based on an intervention procedure performed by a Licensed Nutritionist Doctor for weight loss and loss of fat percentage in patients who need it.

DETAILED DESCRIPTION:
Medical Supervised Duodenal-Enteral Feeding for Overweight, Obesity and Increased Body Fat Percentage Treatment based on an intervention procedure performed by a Licensed Nutritionist Doctor for weight loss and loss of fat percentage in patients who need it. The feeding is by nasogastric-duodenal tube depending on the desired fat loss and / or weight in relation to the basal metabolism. Feeding by tube of 12-29 days, continuing with personalized nutritional treatment for 2 weeks and physical activity during the protocol. Losses of weight and / or expected fat greater than 10%. The results will be compared with bariatric surgery. The main objective is to provide a tool for the obesity epidemic that can be applied worldwide by doctors without the complications of surgery and with a lower price for health systems and controlling the actions of the hormones leptin and ghrelin.

ELIGIBILITY:
Inclusion Criteria:

- Desire for weight loss, desire to improve body image, voluntariness

Exclusion Criteria:

- esophageal alteration or swallowing, not sign the informed consent, acute active disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Weightloss | Change from Baseline weight at 1 and 3 months
  Decrease, minor difference in weight at the end of treatment

SECONDARY OUTCOMES:
Fat loss | Change from Baseline fat percentage at 1 and 3 months
  Decrease, minor difference in percentage of fat at the end of treatment
Loss of measures | Change from Baseline measures at 1 and 3 months
  Decrease of measurements in perimeters (arm, waist, hip, thigh)

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Kuzmar, Dr, Principal Investigator — BiomediKcal - Advanced Medical Nutrition & Lifestyle Center
Locations (1):
- BiomediKcal - Advanced Medical Nutrition & Lifestyle Center, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No
Only available for scientific journal review process

REFERENCES:
- [Result] Kuzmar I, Rizo M, Cortes-Castell E. Adherence to an overweight and obesity treatment: how to motivate a patient? PeerJ. 2014 Jul 29;2:e495. doi: 10.7717/peerj.495. eCollection 2014. PMID 25101227
- [Result] Carey DG, Pliego GJ, Raymond RL, Skau KB. Body composition and metabolic changes following bariatric surgery: effects on fat mass, lean mass and basal metabolic rate. Obes Surg. 2006 Apr;16(4):469-77. doi: 10.1381/096089206776327378. PMID 16608613
- [Result] Carey DG, Pliego GJ, Raymond RL. Body composition and metabolic changes following bariatric surgery: effects on fat mass, lean mass and basal metabolic rate: six months to one-year follow-up. Obes Surg. 2006 Dec;16(12):1602-8. doi: 10.1381/096089206779319347. PMID 17217636
- [Result] Kuzmar I, Cortes E, Rizo M. Age group, menarche and regularity of menstrual cycles as efficiency predictors in the treatment of overweight. Nutr Hosp. 2014 Oct 30;31(2):637-41. doi: 10.3305/nh.2015.31.2.7501. PMID 25617544
- [Result] Strain GW, Gagner M, Inabnet WB, Dakin G, Pomp A. Comparison of effects of gastric bypass and biliopancreatic diversion with duodenal switch on weight loss and body composition 1-2 years after surgery. Surg Obes Relat Dis. 2007 Jan-Feb;3(1):31-6. doi: 10.1016/j.soard.2006.09.002. Epub 2006 Nov 20. PMID 17116424